CLINICAL TRIAL: NCT05470426
Title: Viral Excretion and Its Influencing Factors Among COVID-19 Omicron Recurrence Patients
Brief Title: Viral Excretion Among COVID-19 Omicron Recurrence Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-2022-0102
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: COVID-19 Recurrence; Surface Contamination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: COVID-19 Omicron Recurrence — COVID-19 Omicron Recurrence

SUMMARY:
The study analyzes the viral nucleic acid excretion and its influencing factors of SARS-COV-2 Omicron recurrence patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nucleic acid detection N gene and ORF gene Ct value < 40 after discharge from hospital
* Being able to provide basic information, living habits, vaccination information, admission information

Exclusion Criteria:

* Single gene target positive
* Patients with incomplete baseline data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with COVID-19 Omicron Recurrence
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
COVID-19 Omicron Recurrence | Six months
  COVID-19 Omicron Recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided